CLINICAL TRIAL: NCT05728931
Title: New Biomarkers in Auto-immune Encephalitis and Neurological Paraneoplastic Syndromes
Acronym: DeNobio
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 748
Record Dates: First submitted 2022-11-21; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Paraneoplastic Neurological Syndrome; Autoimmune Encephalitis
Keywords: Paraneoplastic Neurological Syndrome; Autoimmune Encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples (0.5ml), CSF cerebrospinal Fluid (0.2ml), buffy coat (0.5ml), cells or tumors (FFPE block) have been collected in SNP collection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Test of biological samples — Different tests can be use on biological sample : western bloc, dot blot, immune-fluorescence, immunoprecipitation, CBA, functional test, epitope research, IgG title

SUMMARY:
Autoimmune encephalitis (AE) and paraneoplastic neurological syndromes (PNS) are rare neuroimmune syndromes with a wide range of clinical presentation but without pathognomonic clinical sign facilitating the diagnosis. A lot of differential diagnoses are possible such as neurodegenerative diseases or viral infections. Although rare the diagnosis of AE or PNS is essential because despite severe neurological symptoms, patients can be cured by appropriate immunotherapy. Autoantibodies highly specific of AE and PNS has been described in the serum and cerebrospinal fluid of the patients and can be used as biomarkers of the disease. Their presence can predict an autoimmune origin and in many cases a good prognosis after immunotherapy. However, if some autoantibodies are now well-characterized and industrial kits have been developed to detect them, in numerous cases of highly suspect AE or PNS no specific autoantibodies are identified leading frequently to an inappropriate treatment. Furthermore, as the mechanisms of AE and PNS is still unknown, treatments are not optimal and in some cases inefficient. There is no prognosis biomarker able to predict the patient's sensitivity to immunotherapy and there are only few clues to know how the immune system can provoke the neuropsychiatric symptoms observed in the patients. The investigators will use this project to better characterize AE and PNS patients to identify new diagnostic and prognostic biomarkers and develop new diagnostic tools.

ELIGIBILITY:
* Inclusion Criteria * :

  * patient with neurological disorder
  * patient without antibody
* Exclusion Criteria * :

  * patient with characterized antibody
  * patient without neurological disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient without antibodies known with neurological disorder and include in biobank of "centre de reference des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes".
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2032-01-15 (Estimated)

PRIMARY OUTCOMES:
Description of new biomarkers | Baseline
  Results of diagnostics tests for each patient, description of marking

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites autoimmunes, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided